CLINICAL TRIAL: NCT00852358
Title: A Study of Intrathecal Enzyme Replacement for Cognitive Decline in Mucopolysaccharidosis I
Brief Title: A Study of Intrathecal Enzyme Therapy for Cognitive Decline in MPS I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patricia I. Dickson, M.D. (Individual)
Collaborators: The Ryan Foundation (Other); BioMarin Pharmaceutical (Industry); Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Minnesota (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor-Investigator, Patricia I. Dickson, M.D., Associate Professor of Pediatrics, Dickson, Patricia I., M.D.
Organization: Dickson, Patricia I., M.D. (Individual)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MIRC-002; MIRC-002; IRB Project No. 13270-01; IND 104,354; U54NS065768 (NIH)
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Cognitive Decline; Mucopolysaccharidosis I; Hurler-Scheie Syndrome; Scheie Syndrome; Lysosomal Storage Disease
Keywords: mucopolysaccharidosis; Hurler-Scheie; Scheie; laronidase; cognitive decline; central nervous system; enzyme replacement therapy; intrathecal; LA Biomed
MeSH Terms: conditions — Cognitive Dysfunction; Mucopolysaccharidosis I; Lysosomal Storage Diseases; Mucopolysaccharidoses | interventions — Iduronidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intrathecal laronidase (Experimental): The Experimental treatment group will receive study assessments and intrathecal laronidase (1.74 mg laronidase) treatments every 1-3 months beginning at start of study.
  Interventions: Drug: laronidase
- Control Group (Other): During the first 11 months, the control group will receive study assessments but will be unblinded with no intrathecal treatment or placebo administered. Beginning at month 12, the control group will receive intrathecal laronidase (1.74 mg) treatment every 3 months (months 12, 15, 18, and 21).
  Interventions: Drug: laronidase

INTERVENTIONS:
Drug: laronidase — For the treatment group, intrathecal rhIDU injections will consist of 3 cc of Aldurazyme® (laronidase) (approximately 1.74 mg) diluted with 6 cc of Elliotts B® solution for a total injection of 9 cc. The diluted enzyme will be administered via a lumbar puncture (IT) on day 0 after baseline assessments. IT injections will be repeated on days 30, 60, and 90. The subsequent doses will be administered at 3-month intervals for a total of 10 doses during the two-year period. Control patients will not receive treatment, lumbar puncture, or placebo, but will undergo all other study procedures and assessments during year one. Control patients will then enter a treatment phase consisting of four IT doses at 3-month intervals.
  Other Names: Aldurazyme; recombinant human alpha-l-iduronidase

SUMMARY:
This is a 24-month study of the use of laronidase administered into the spinal fluid to treat cognitive decline in mucopolysaccharidosis I (MPS I). MPS I is a rare genetic condition due to deficiency of the enzyme alpha-l-iduronidase. Laronidase is the manufactured form of the enzyme alpha-l-iduronidase.

MPS I is a heterogeneous disease with several clinical phenotypes ranging from the most severe, Hurler syndrome, to the attenuated forms, Hurler-Scheie and Scheie. Although patients with milder forms of MPS I may not have grossly observable problems with cognition, these patients do have learning difficulties that are apparent in school and with neuropsychological testing. The goal of this study is to evaluate whether intrathecal recombinant human alpha-l-iduronidase (rhIDU) injections can stabilize or improve cognitive decline in individuals with MPS I.

DETAILED DESCRIPTION:
This study is a 24-month open label, prospective, randomized trial in 16 MPS I patients age six years or older who have documented evidence of cognitive decline. The study will test the safety and efficacy of intrathecal recombinant human alpha-L iduronidase (rhIDU) to reduce or stabilize cognitive decline by assessing the subjects at baseline with neuropsychological, clinical, radiological, and biochemical evaluations and then monitoring the change in these parameters during a regimen of first monthly, then quarterly, intrathecal treatments with rhIDU. The clinical safety of the regimen will be assessed by monitoring of adverse events, cerebrospinal fluid (CSF) laboratory assessments, and clinical evaluations.

Subjects will be randomized to a treatment or a control group for 12 months, following which all subjects will receive 12 months of active treatment. During the first 12 months, the control group will receive similar study assessments but will be unblinded with no placebo administered. Subjects will have extensive baseline screening evaluations, after which subjects who were randomized to the treatment group will receive their first dose of intrathecal rhIDU. The enzyme will be administered via intrathecal injection at 1-3 month intervals throughout the 24-month study period. There will be a mid-study analysis after 12 months comparing changes in IQ and memory tests between controls and the treatment group. If pre-established criteria of improvement are met, the study will terminate at the 12 month point. If shown to be effective, intrathecal enzyme replacement therapy (ERT) would be the only treatment for cognitive decline in patients who do not qualify for and/or are unable to have hematopoietic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* The presence of MPS I disease as documented by low α-L-iduronidase activity
* Age six years or older.
* The presence of acquired cognitive deficits as demonstrated by:

  1. A score of one standard deviation below mean on IQ testing or in one domain of neuropsychological function (language, memory, or non-verbal ability), OR
  2. Documented historical evidence of a decline of greater than one standard deviation on sequential testing, OR
  3. A score between 0.75 and 1 standard deviation below the mean, AND the cognitive deficit affects daily performance.
* The decline in function is not explainable by other neurological or psychiatric factors.
* Subject and/or guardian willing and able to provide written informed consent.
* Negative urine pregnancy test at screening (non-sterile females of child-bearing potential only)
* Currently using two acceptable methods of birth control as determined by the investigator and willing to continue to use acceptable birth control during their participation in the study (non-sterile females of child-bearing potential who are sexually active only)
* Willing and able to comply with study procedures. For example, the subjects must be able to complete written and computer-based testing. The subjects must be able to lie still in the MRI scanner for at least 40 minutes without sedation.

Exclusion Criteria:

* The subject has undergone hematopoietic stem cell transplantation
* Recent initiation of intravenous Aldurazyme® therapy with less than 6 months of therapy. Subjects who have been receiving Aldurazyme® therapy for more than 6 months, and those who have never received Aldurazyme® therapy, will be allowed to enroll
* Pregnant or lactating, or considering pregnancy
* Receipt of an investigational drug or procedure within 30 days of enrollment
* A condition, medical or other, that prevents participation in the study, including severe auditory or visual impairment, significant lumbar pathology, lumbar catheter, or recent major surgery within 6 weeks that would preclude their ability to participate.
* Infusion reactions to intravenous Aldurazyme® therapy that require ongoing medical intervention, special prophylaxis or altered rate or dose of enzyme administration
* The subject has a programmable VP shunt that is incompatible with the 3 Tesla MRI magnet and is unable or unwilling to undergo shunt revision to a MRI compatible device.
* The subject has another contraindication for MRI, such as nonremovable metal in the body.
* The subject has severely impaired spinal CSF flow, demonstrated by failure of appearance of 99mTechnetium-DTPA in the basal cisterns by 4 hours after intra-lumbar administration.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to assess the ability of intrathecal α-L-iduronidase to be administered safely | 24 months

SECONDARY OUTCOMES:
The objective of this study is to assess the ability of intrathecal α-L-iduronidase to stabilize or reverse cognitive decline. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Chen, MD, Principal Investigator — Los Angeles Biomedical Institute at Harbor-UCLA; Patricia I Dickson, MD, Principal Investigator — Los Angeles Biomedical Institute at Harbor-UCLA
Locations (3):
- United States (3):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Los Angeles Biomedical Institute at Harbor-UCLA, Torrance, California
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No